CLINICAL TRIAL: NCT04604730
Title: Role of Protective Stoma After Primary Anastomosis for Generalized Peritonitis Due to Perforated Diverticulitis: a Prospective Multicenter Randomized Trial
Brief Title: Role of Protective Stoma After Primary Anastomosis for Generalized Peritonitis Due to Perforated Diverticulitis
Acronym: DIVERTI2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/0409/HP
Record Dates: First submitted 2020-10-15; First posted 2020-10-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Peritonitis
Keywords: peritonitis; perforated diverticulitis; primary anastomosis; protective stoma
MeSH Terms: conditions — Peritonitis | interventions — Anastomosis, Surgical

STUDY DESIGN:
Intervention Model Description: Sequential assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary anastomosis without protective stoma (Experimental): Primary anastomosis without protective stoma
  Interventions: Procedure: Primary anastomosis without protective stoma
- Anastomosis with protective stoma (Active Comparator): Anastomosis with protective stoma
  Interventions: Procedure: Anastomosis with protective stoma

INTERVENTIONS:
Procedure: Primary anastomosis without protective stoma — Primary anastomosis without protective stoma
  Arms: Primary anastomosis without protective stoma
Procedure: Anastomosis with protective stoma — Anastomosis with protective stoma
  Arms: Anastomosis with protective stoma

SUMMARY:
This study is designed to be a multicentre, prospective, comparative, randomised trial, evaluating the efficacy of two surgical strategies for the treatment of generalised peritonitis due to perforated diverticulitis. Results will be analysed according to an intention to treat principle (after selection and patient consent). Immediately before surgery, the patient will be randomly assigned to sigmoidectomy with primary anastomosis or to sigmoidectomy with primary anastomosis and diverting stoma. Sigmoidectomy will be performed through a midline laparotomy or laparoscopically according to the standard technique. In the control arm, a protective stoma will be performed at the end of surgery. A stoma reversal operation will be performed at least 3 months after the first operation and after performing a cologram by water soluble contrast between 4 and 8 weeks to check for the absence of fistula or stenosis at the level of the anastomosis. Stoma reversal will be performed with a trephine incision.

Post-stoma closure follow-ups will be planned and all morbidity/mortality will be recorded. All patients will be examined at 6, 12, and 24 weeks after the initial surgery, in the surgical department where they were operated; a final study visit will be carried out 12 months (evaluation of primary endpoint) after surgery. The parameters explored at medical examinations will be: • Occurrence of complications • Quality of life assessment

DETAILED DESCRIPTION:
This study is designed to be a multicentre, prospective, comparative, randomised trial, evaluating the efficacy of two surgical strategies for the treatment of generalised peritonitis due to perforated diverticulitis. Results will be analysed according to an intention to treat principle. The diagnosis will be established by the surgeon investigator on clinical data, imagery and operative findings during a laparotomy or laparoscopy. After selection and patient consent and immediately before surgery, the patient will be randomly assigned to sigmoidectomy with primary anastomosis or to sigmoidectomy with primary anastomosis and diverting stoma. Sigmoidectomy will be performed through a midline laparotomy or laparoscopically according to the standard technique, with lateral to medial mobilisation of the left colon, mobilisation of splenic flexure and identification of left ureter. The rectosigmoid junction will be exposed and transected with a stapler. Proximal section will be performed on a healthy colonic segment. The anastomosis will be performed according to the surgeon investigator's preference (mechanical or manual anastomosis; end to end or side to end).

Decisions to clean the colon intraoperatively and to place a drain will be left to the surgeon's discretion. In the control arm, a protective stoma will be performed at the end of surgery. A stoma reversal operation will be performed at least 3 months after the first operation and after performing a cologram by water soluble contrast between 4 and 8 weeks to check for the absence of fistula or stenosis at the level of the anastomosis. Stoma reversal will be performed with a trephine incision.

Post-stoma closure follow-ups will be planned and all morbidity/mortality will be recorded. All patients will be examined at 6, 12, and 24 weeks after the initial surgery, in the surgical department where they were operated; a final study visit will be carried out 12 months (evaluation of primary endpoint) after surgery. The parameters explored at medical examinations will be: • Occurrence of complications • Quality of life assessment

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients operated for purulent or fecal peritonitis (Hinchey grade III and IV) secondary to perforated diverticulitis of the left colon and treated by resection with primary anastomosis
3. Person informed and having signed his consent. If the patient is unable to sign his consent, the consent will be signed by his representative ((1) the trusted person, or failing that, (2) a family member, or (3) a relative of the person concerned) (Article L1122-1-1 of the CSP). In this case, consent to continue the study will subsequently be requested from the patient. --> In addition, due to the vital urgency represented by hospitalisation in intensive care for purulent or fecal peritonitis, inclusion without prior collection of the consent of the patient or his/her representative is possible in the case where the patient is not capable of giving consent and his/her representative is not present at the time of inclusion (Article L1122-1-3 of the CSP). In this case, the patient or his/her representative will be informed as soon as possible and his/her written consent will be requested for the possible continuation of this research and the use of the data concerning him/her.
4. Patient able to comply with the study protocol, in the investigator's judgment
5. Patient affiliated with, or beneficiary of a social security (health insurance) category

Non-inclusion Criteria:

1. Physical states that prevent patient participation (e.g. septic shock or multivisceral failure)
2. Steroid treatment > 20 mg daily
3. Prior pelvic irradiation
4. Immunocompromised status
5. Known progressive cancer
6. American Society of Anesthesiologists grade IV
7. Peritonitis secondary to perforated diverticulitis of the right colon
8. Patient is a pregnant (positive blood pregnancy test) or breastfeeding (lactating) woman or intending to become pregnant during the study
9. Person deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision)
10. Simultaneous participation in another interventional research

Exclusion Criteria:

1. Failure to obtain the consent of the patient or the patient's representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of overall morbidity between "with protective stoma" and "without protective stoma" | 12 months posteoperatively
  Overall morbidity graded 0 to 5 according to the Clavien-Dindo classification All complications occurring during hospitalization will be collected. Late complications occurring after hospitalization will be collected during follow-up.

SECONDARY OUTCOMES:
Comparison of the rate of death between "with protective stoma" and "without protective stoma" | 3 months postoperatively
  rate of death at 3 months after surgery (%)
Comparison of the rate of reinterventions between "with protective stoma" and "without protective stoma" | 12 months postoperatively
  the rate of reinterventions after the surgery (%)
Comparison of the rate of incisional surgical site infection (SSI) between "with protective stoma" and "without protective stoma" | 12 months postoperatively
  the rate of incisional SSI (%)
Comparison of the rate of organ/space SSI between "with protective stoma" and "without protective stoma" | 12 months postoperatively
  the rate of organ/space SSI (%)
Comparison of the rate of wound disruptions between "with protective stoma" and "without protective stoma" | 12 months postoperatively
  the rate of wound disruptions (%)
Comparison of the rate of anastomotic leaks between "with protective stoma" and "without protective stoma" | 12 months postoperatively
  the rate of anastomotic leaks (%)
Comparison of operating time between "with protective stoma" and "without protective stoma" | surgery
  time of surgery (hours)
Comparison of length of postoperative hospital stay between "with protective stoma" and "without protective stoma" | 6 months postoperatively
  Length of postoperative hospital stay (days)
Comparison of Intensive Care Unit (ICU) length of stay between "with protective stoma" and "without protective stoma" | 6 months postoperatively
  ICU length of stay (days)
Comparison of the number of patients alive without stoma between "with protective stoma" and "without protective stoma" | 12 months after initial surgery
  Number of patients alive without stoma at 12 months after initial surgery
Comparison of the quality of life between "with protective stoma" and "without protective stoma" | 6, 12, 26 and 52 weeks after primary surgery
  Quality of life evaluated using the Short Form Health Survey (SF-36) questionnaire at baseline, 6, 12, 26 and 52 weeks after primary surgery Score from 1 to 30
Comparison of the quality of life between "with protective stoma" and "without protective stoma" with "EuroQol-5 Dimensions" questionnaire | 6, 12, 26 and 52 weeks after primary surgery
  Quality of life evaluated using EuroQol-5 Dimensions (EQ-5D) questionnaire at baseline, 6, 12, 26 and 52 weeks after primary surgery Each dimension has three levels of response: no problems (coded 1), some problems (coded 2) and major problems (coded 3), which defines 243 possible health states (35), to which can be added unconscious and dead states, for a total of 245 states. Thus, the health states range from "11111" (no problems on all dimensions) to "33333": major problems on all dimensions + visual analog scale from 0 to 100, 0 being the worst and 100 the best
Comparison of the quality of life between "with protective stoma" and "without protective stoma" with the Gastrintestinal Quality of Life Index questionnaire | 6, 12, 26 and 52 weeks after primary surgery
  Quality of life evaluated using Ethe Gastrintestinal Quality of Life Index questionnaire at baseline, 6, 12, 26 and 52 weeks after primary surgery Score from 0 to 144, the higher the score, the better the quality of life
Comparison of the cost utility between "with protective stoma" and "without protective stoma" | 12 months after primary surgery
  Quality-Adjusted Life Year (QALY) derived from the EQ5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BRIDOUX, Pr, Principal Investigator — University Hospital, Rouen
Locations (20):
- France (20):
  - CHR Beauvais, Beauvais, Beauvais
  - CHU Amiens, Amiens
  - CH Beauvais, Beauvais
  - CHU Besançon, Besançon
  - APHP Avicenne, Bobigny
  - CHU Brest, Brest
  - CHU Caen, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - APHP Henri Mondor, Créteil
  - CHU Grenoble, Grenoble
  - CHU Limoges, Limoges
  - CHU Lyon, Lyon
  - APHM Hôpital Nord, Marseille
  - APHM La Timone, Marseille
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nimes, Nîmes
  - APHP St Antoine, Paris
  - CHU Rouen, Rouen
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinson J, Tuech JJ, Ouaissi M, Mathonnet M, Mauvais F, Houivet E, Lacroix E, Rondeaux J, Sabbagh C, Bridoux V. Role of protective stoma after primary anastomosis for generalized peritonitis due to perforated diverticulitis-DIVERTI 2 (a prospective multicenter randomized trial): rationale and design (nct04604730). BMC Surg. 2022 May 16;22(1):191. doi: 10.1186/s12893-022-01589-w. PMID 35578267